CLINICAL TRIAL: NCT06376643
Title: Evaluation of an Augmented Reality and Screen-based Decision Support System for Cardiopulmonary Arrest: a Multicenter, Randomized Clinical Trial
Brief Title: Augmented Reality to Support Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johan Siebert, MD (Other)
Collaborators: University Hospital, Geneva (Other); Alberta Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Johan Siebert, MD, MD, PD, Deputy Head, Pediatric Clinical Research Platform
Organization: Pediatric Clinical Research Platform (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: InterFACE-AR
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cardiopulmonary Arrest; Resuscitation; Pediatric
Keywords: Cardiopulmonary Resuscitation; Augmented Reality; Digital Health; Pediatrics
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Open-label, prospective, multicenter, cluster randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to blind study participants to study arm allocation due to the nature of the intervention(s), but they will be blinded to study objectives. The statistician will be blinded regarding the allocation of participants to the study arms for results analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Augmented Reality) (Experimental): Participants that will use the augmented reality supportive tool during the simulation-based pediatric scenario.
  Interventions: Device: Augmented reality supportive tool
- Arm B (Conventional methods) (Active Comparator): Participants that will use conventional methods during the simulation-based pediatric scenario.
  Interventions: Other: Conventional method (AHA pocket reference card)

INTERVENTIONS:
Device: Augmented reality supportive tool — Participants will view a standardized orientation video describing the clinical environment, equipment, manikin functionality, and participant roles, followed by a 15-minute table-top practice simulation where participants have opportunity to use the assigned intervention by running through a cardiac arrest scenario.
  Then, participants will undertake a 20-minute tightly standardized cardiac arrest simulation scenario using a high-fidelity pediatric manikin. The scenarios will be videotaped from a bird's-eye view angle at the foot of the bed, along with three action video cameras worn by the participants, and positioned within the room.
  Following completion of the scenario, participants will fill out five surveys (see secondary outcomes), which together take about 15 minutes to fill.
  Arms: Arm A (Augmented Reality)
Other: Conventional method (AHA pocket reference card) — Participants will view a standardized orientation video describing the clinical environment, equipment, manikin functionality, and participant roles, followed by a 15-minute table-top practice simulation where participants have opportunity to use the assigned intervention by running through a cardiac arrest scenario
  Then, participants will undertake a 20-minute tightly standardized cardiac arrest simulation scenario using a high-fidelity pediatric manikin. The scenarios will be videotaped from a bird's-eye view angle at the foot of the bed, along with three action video cameras worn by the participants, and positioned within the room.
  Following completion of the scenario, participants will fill out five surveys (see secondary outcomes), which together take about 15 minutes to fill.
  Arms: Arm B (Conventional methods)

SUMMARY:
A prospective, multicenter, randomized clinical trial in two tertiary pediatric emergency department. It will assess, amongst pediatric healthcare teams, whether the use of augmented reality supportive devices improves adherence to American Heart Association (AHA) advanced life support guidelines and performance, while reducing medication errors, when compared to groups using the AHA pocket reference card (control) during standardized, simulation-based, pediatric in-hospital cardiac arrest (IHCA) scenarios. Seventy participants will be randomized. The primary endpoint is the time to first dose of epinephrine.

DETAILED DESCRIPTION:
Each year, thousands of children experience cardiopulmonary arrests (CA), requiring immediate and accurate resuscitation for favorable outcomes. However, adherence to American Heart Association (AHA) advanced life support guidelines remains suboptimal, hindered by cognitive and communication challenges in high-stress cardiopulmonary resuscitation (CPR) situations. To address this problem, will assess a novel augmented reality (AR)-assisted digital health solution designed to offer personalized, real-time decision support for team leaders and medication nurses, while concurrently optimizing team situational awareness and communication by projecting a dynamic care roadmap onto a large screen in the resuscitation room, controlled via a mobile tablet app.

The solution comprises three essential digitally interconnected elements: 1) a mobile app that presents clinical algorithms alongside patient data, guiding the resuscitation team through step-by-step procedures, 2) a giant screen that displays real-time patient information and task progress for the entire resuscitation team, and 3) augmented reality devices worn by team members, providing role-specific guidance and decision support based on data collected by the app.

In this trial, we will assess, amongst pediatric healthcare teams, whether the use of the AR-assisted tool improves adherence to AHA resuscitation guidelines and performance, while reducing medication errors, when compared to groups using the AHA pocket reference card (control) in an open-label, prospective, multicenter, cluster randomized (1:1 ratio) clinical trial. Sixty physicians and nurses will be recruited to form teams of 7, each managing simulated pediatric in-hospital cardiac arrest (IHCA) scenarios using either an AR-assisted tool or conventional AHA pocket reference cards. Each team will comprise three participants assigned to the roles of 1) Team Leader (a physician), 2) Charting Nurse, and 3) Medication Nurse, with two CPR Providers, an Airway Provider, and a Bedside Provider roles filled by research actors. All participants and actors will view a CPR Coach orientation video to ensure understanding of the CPR Coach and Provider functions

The primary outcome is the time in seconds to first dose of epinephrine. Secondary outcomes are times to CPR initiation, defibrillation, drug delivery, airway securing, the rate of medication errors, CPR pause frequency, CPR quality (excellent CPR percentage, chest compression fraction, peri-shock pause duration), provider workload (NASA-TLX survey) and stress (STAI), user experience (UEQ), system usability (SUS), and technology acceptance (UTAUT).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the team leader include: attending physician, fellow, or senior resident in emergency medicine, pediatric emergency medicine, pediatrics, pediatric critical care, or pediatric anesthesia.
* Inclusion criteria for the medication and charting nurse roles include: nurse in pediatric emergency medicine, general pediatrics, or other pediatric acute care specialty.
* Inclusion criteria for all other team members include: pediatric attending physician, resident, fellow, nurse or respiratory therapist.
* Participants must have prior basic life support training.
* Participation agreement.

Exclusion Criteria:

* Decline to provide informed consent
* Previously enrolled
* Unable to perform tasks required of the role

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Time to first dose of epinephrine | 20 minutes
  The primary outcome is the time in seconds to first dose of epinephrine administration

SECONDARY OUTCOMES:
Time to initiation of cardiopulmonary resuscitation | 20 minutes
  The time in seconds from the investigator's clinical statement to initiation of chest compression
Time to defibrillation | 20 minutes
  The time in seconds from the investigator's clinical statement to each manual defibrillator shock delivery
Time to delivery of epinephrine | 20 minutes
  The time in seconds from the investigator's clinical statement to intravenous injection of epinephrine to treat underlying condition
Time to delivery of amiodarone | 20 minutes
  The time in seconds from the investigator's clinical statement to intravenous injection of amiodarone to treat underlying condition
Time to secure definitive airway | 20 minutes
  The time in seconds from the investigator's clinical statement to the successful establishment of a definitive airway via endotracheal intubation
Medication dosage errors | 20 minutes
  Errors in drug dose administration (milligrams), defined as a deviation from the correct weight-based dose of more than 10% according to predefined, expert consensus-based criteria, will be measured (i.e., absolute and percentage deviation) in each allocation group as a deviation from the 2020 AHA Pediatric Advanced Life Support cardiac arrest algorithm.
Types of Medication Errors | 20 minutes
  The nature of the error type will be recorded, such as incorrect drug selection (i.e., administering the wrong medication), administration timing errors (i.e., administering the medication at the wrong time during the resuscitation process), labeling errors (i.e., misinterpreting or misreading the medication label), equipment-related errors (i.e., issues related to the functioning or availability of equipment needed for drug administration [e.g., syringe malfunction]), and documentation errors (i.e., inaccurate or incomplete recording of medication administration details)
Frequency of Medication Errors | 20 minutes
  Number of times medication errors occur during the cardiac arrest scenario
Frequency of pauses in cardiopulmonary resuscitation | 20 minutes
  Number of times of cardiopulmonary resuscitation pauses during the cardiac arrest scenario
Duration of pauses in cardiopulmonary resuscitation | 20 minutes
  The total time in seconds of cardiopulmonary resuscitation pauses during the cardiac arrest scenario
Causes of pauses in cardiopulmonary resuscitation | 20 minutes
  The causes leading to resuscitation interruptions will be identified and documented
Cardiopulmonary resuscitation quality: Percentage of overall excellent cardiopulmonary resuscitation | 20 minutes
  The proportion of cardiopulmonary resuscitation administrations that meet the predefined AHA standards for high-quality resuscitation techniques.
Cardiopulmonary resuscitation quality: Chest compression fraction | 20 minutes
  The fraction of time in seconds that chest compressions are being performed over the total cardiopulmonary resuscitation duration
Cardiopulmonary resuscitation quality: Peri-shock pause duration | 20 minutes
  The length of time in seconds between the cessation of chest compressions and the delivery of a defibrillation shock during cardiopulmonary resuscitation
Provider workload (NASA-TLX) | 15 minutes
  Assessed via NASA-TLX. It measures mental burden across 6 dimensions: mental, physical, temporal demands, performance, effort, and frustration. Scores range from 0 to 100 in 5-point increments (0: no task load; 100: maximal task load). Participants rate each dimension based on their perceived workload. To combine the dimensions into a final score, a weighting procedure is used. This involves comparing each dimension with every other dimension to determine its relative importance in influencing workload. Participants select the dimension that contributes most to workload in each pair of comparisons. Each dimension is then weighted based on the participant's selections, with higher weights given to dimensions that are chosen more frequently. The weighted scores for each dimension are summed to calculate the overall score, which ranges from 0 (minimal task load) to 100 (maximal task load)
User Experience Questionnaire (UEQ) | 15 minutes
  UEQ is a widely used questionnaire to measure the subjective impression of users towards the user experience of products. The UEQ is a semantic differential with 26 items that are grouped into six scales (Attractiveness, Perspicuity, Efficiency, Dependability, Stimulation, and Novelty). Each scale represents a distinct usability quality aspect. The minimum value is 0 (i.e., the worst user experience) and the maximum value is 100 (i.e., the best user experience). Participants will be asked to complete the UEQ directly after they have completed the resuscitation scenario
System Usability Scale (SUS) | 15 minutes
  SUS is a widely used questionnaire for assessing the perceived usability of a system or product. The SUS consists of a 10-item questionnaire where users rate their agreement or disagreement with a series of statements regarding the usability of a system using a 5-point Likert scale (1 to 5). The minimum value is 0 (i.e., the system is not usable) and the maximum value is 100 (i.e., the system is absolutely usable). Participants will be asked to complete the SUS directly after they have completed the resuscitation scenario
Unified Theory of Acceptance and Use of Technology questionnaire (UTAUT) | 15 minutes
  The UTAUT consists of eight domains (performance expectancy, effort expectancy, social influence, facilitating conditions, hedonic motivation, price value, habit, and behavioural intention). This measure will be adapted to assess participants' perceived usability, usefulness, and intention to use the augmented reality-aided tool after study completion. Responses are rated on a 7-point likert scale from 1=Strongly disagree to 7=Strongly agree. Participants will be asked to complete the UTAUT directly after they have completed the resuscitation scenario
State-Trait Anxiety Inventory (STAI) form Y-1 | 15 minutes
  This questionnaire is composed of 20-item self-report subscales to measure the temporary state of anxiety at the time of reporting (STAI form Y-1), which can be affected by stressful situations. Each item is answered on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much). After reversing the scores for stress-absent items (ie, items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20), the total score is calculated by summing up the weighted scores for the 20 items. STAI ranges from 20 to 80, with higher scores being positively correlated with greater stress. The range of possible scores range from a minimum score of 20 to a maximum score of 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80). Participants will be asked to complete the STAI directly after they have completed the resuscitation scenario
Visual attention patterns of team leader and medication nurse on augmented reality and resuscitation room elements | 20 minutes
  Duration and number of visual fixations on pre-defined area of interest (AOI) for the team leader and medication nurse, as captured by the augmented reality device (Microsoft Hololens2). AOIs will include the holograms projected within each augmented reality device, as well as the LCD screen within the resuscitation room and manikin for the team leader.
Team Emergency Assessment Measure (TEAM) survey | 10 minutes
  The TEAM survey is a validated tool designed to assess team performance during emergency scenarios, focusing on non-technical skills. It consists of 11 items rated on a 5-point Likert scale (0 [Never/Hardly ever] to 4 [Always/Nearly always]) across three domains: Leadership, Teamwork, and Task Management, with an additional overall performance rating. Scores range from 0 (poor performance) to 44 (excellent performance), providing a comprehensive measure of team dynamics, communication, and coordination. Participants will complete the TEAM survey immediately after each resuscitation scenario to evaluate the team's effectiveness in managing the simulated IHCA
Concise Assessment of Leader Management (CALM) Survey | 10
  The CALM survey is a validated tool for assessing leadership in acute resuscitation scenarios, focusing on the Team Leader's performance. It includes 15 four-point Likert scale items (rarely, sometimes, mostly, always) across 4 domains-Leadership (role and style, 2 items), Communication (clarity and closed-loop reinforcement, 2 items), Team Management (role assignment, task direction, workload balance, team engagement, and case summarization, 5 items), and Medical Management (task prioritization, global awareness, patient reassessment, care planning, and help-seeking, 5 items)-plus 1 dichotomous behavioral item (yes/no on role announcement) and 1 global rating item comparing the leader to peers (below expected, as expected, above expected, top 5%). Scores for the Likert items range from 15 (poor leadership) to 60 (outstanding leadership), with additional binary and comparative assessments. Team members will complete the CALM survey immediately after each resuscitation scenario.

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Siebert, MD, PD, Principal Investigator — Geneva Children's Hospital, Geneva, Switzerland; Adam Cheng, Prof, Study Director — Alberta Children's Hospital, Calgary, Canada
Locations (2):
- Alberta Children's Hospital, Calgary, Alberta, Canada
- Geneva Children's Hospital, Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No